CLINICAL TRIAL: NCT01082614
Title: Evaluation of the Use of Arterial Pulse Waveform Contour Analysis for Early Goal Directed Therapy in Patients Undergoing Major Abdominal Surgery
Brief Title: Arterial Pulse Waveform Contour Analysis for Intraoperative Goal Directed Therapy in Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59162
Record Dates: First submitted 2010-03-03; First posted 2010-03-08 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard fluid management (No Intervention): standard intraoperative fluid management as determined by usual monitoring and decision making applied by anesthesiology team
- Goal directed therapy (Experimental): Intraoperative fluid management guided by stroke volume variation determined by arterial pressure pulse wave contour analysis
  Interventions: Device: Vigileo

INTERVENTIONS:
Device: Vigileo — Pulse contour waveform analysis derived stroke volume variation will be used to guide intraoperative fluid administration. Additional fluid boluses will be given to the patient when SVV > 12%.
  Other Names: Vigileo model number MHM1
  Arms: Goal directed therapy

SUMMARY:
This study evaluates whether using information from a special arterial blood pressure monitor to guide how much fluid is given during surgery changes how long a patient stays in the hospital after the surgery. There is scientific evidence from using similar information from different devices that this technique might allow us to do a better job giving fluids during surgery and that this may be associated with shorter hospital stay after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring elective or semi-elective major abdominal surgery will be assessed for eligibility.

Exclusion Criteria:

* Age under 18 years old,
* Coagulopathy,
* Significant renal/hepatic dysfunction (creatine >50% or liver enzymes > 50% of normal values),
* Congestive heart failure,
* Cardiac arrhythmias producing irregular rhythms, and
* Patient choice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Applegate II, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Fluid Management | Goal Directed Therapy
Started | 23 | 23
Completed | 20 | 18
Not Completed | 3 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Equipment Malfunction | 0 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Fluid Management | Goal Directed Therapy | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 13 | 21
  >=65 years | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (15.8) | 53.5 (16.2) | 58.95 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Length of Postoperative Hospital Stay
Description: time in days from end of surgery to hospital discharge
Time Frame: within one month
Measure: Mean (Full Range); unit: Days
Arm/Group | Standard Fluid Management | Goal Directed Therapy
Number analyzed (Participants) | 20 | 18
Days | 7.5 [5.25 to 10.75] | 5.0 [3.75 to 8.25]

2. Secondary Outcome: Quality of Recovery Score on Postoperative Day 2
Description: Measure of quality of recovery (QOR) using scoring system in 9 domains as assessed by patient and nursing team. Score for each domain is assigned as 0, 1 or 2; the sum of scores is the QOR score with a range of 0 to 18. Higher scores indicate better quality of recovery after surgery.
Time Frame: Postoperative day 2
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Fluid Management | Goal Directed Therapy
Number analyzed (Participants) | 20 | 18
units on a scale | 15.0 [14.0 to 15.75] | 16.0 [14.75 to 17.0]

3. Secondary Outcome: Quality of Recovery Score on Postoperative Day 4
Description: Measure of quality of recovery (QOR) using scoring system in 9 domains as assessed by patient and nursing team. Score for each domain is assigned as 0, 1 or 2; the sum of scores is the QOR score with a range of 0 to 18. Higher scores indicate better quality of recovery following surgery.
Time Frame: Postoperative day 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Fluid Management | Goal Directed Therapy
Number analyzed (Participants) | 20 | 18
units on a scale | 16.5 [15.0 to 18.0] | 18.0 [17.0 to 18.0]

ADVERSE EVENTS:
Arm/Group | Standard Fluid Management | Goal Directed Therapy
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes